CLINICAL TRIAL: NCT03195543
Title: Assessment of Blood Coagulation Disorders in Patients With Pulmonary Arterial Hypertension and Chronic Thromboembolic Pulmonary Hypertension.
Brief Title: Assessment of Blood Coagulation Disorders in Patients With Pulmonary Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Eleni Vrigkou, PhD candidate, National and Kapodistrian University of Athens
Other Study IDs: ΕΒΔ410/17-9-14
Record Dates: First submitted 2017-06-08; First posted 2017-06-22 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Pulmonary Artery Hypertension; Chronic Thromboembolic Pulmonary Hypertension
Keywords: Blood coagulation disorders; Platelets; Thrombin; Treatment
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Blood Coagulation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with PAH: Diagnostic tests will be performed on patients with Pulmonary Artery Hypertension in order to assess any blood coagulation disorders. Platelet function, coagulation and fibrinolysis will be evaluated by platelet function analyzer-100 (PFA-100), light transmission aggregometry, rotational thromboelastometry (ROTEM) and endogenous thrombin potential.
  Interventions: Diagnostic Test: Platelet function analyzer-100; Diagnostic Test: Light transmission aggregometry; Diagnostic Test: Rotational thromboelastometry; Diagnostic Test: Endogenous thrombin potential
- Patients with CTEPH: Diagnostic tests will be performed on patients with Chronic Thromboembolic Pulmonary Hypertension in order to assess any blood coagulation disorders. Platelet function, coagulation and fibrinolysis will be evaluated by platelet function analyzer-100 (PFA-100), light transmission aggregometry, rotational thromboelastometry (ROTEM) and endogenous thrombin potential.
  Interventions: Diagnostic Test: Platelet function analyzer-100; Diagnostic Test: Light transmission aggregometry; Diagnostic Test: Rotational thromboelastometry; Diagnostic Test: Endogenous thrombin potential

INTERVENTIONS:
Diagnostic Test: Platelet function analyzer-100 — The PFA-100 system evaluates primary hemostasis in whole blood samples.
  Other Names: PFA-100
Diagnostic Test: Light transmission aggregometry — Light transmission aggregometry is the gold standard method for assessing platelet function.
Diagnostic Test: Rotational thromboelastometry — ROTEM is a viscoelastic method for hemostasis testing in whole blood.This assay investigates the interaction of blood cells, coagulation factors and their inhibitors during clotting and subsequent fibrinolysis.
  Other Names: ROTEM
Diagnostic Test: Endogenous thrombin potential — The endogenous thrombin potential assesses the amount of thrombin which can be generated after the in vitro activation of coagulation and represents the balance between pro- and anti-coagulant forces in plasma.
  Other Names: ETP

SUMMARY:
The objective of the present study is to assess blood coagulation disorders in patients with Pulmonary Arterial Hypertension and Chronic Thromboembolic Pulmonary Hypertension. The investigators aim to evaluate any possible coagulation abnormalities related to the patients' primary disease and any possible effects the pulmonary hypertension- specific therapy may have on hemostasis.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a chronic, progressive, pulmonary vascular disease with a multifactorial etiology and a not fully elucidated pathophysiological background. There is a complex and not adequately understood association between PH and the coagulation process.

The aim of the present study is to evaluate hemostasis in patients with PH classified as category 1 of the World Health Organization Pulmonary Hypertension Group (Pulmonary Arterial Hypertension, PAH) and 4 (Chronic Thromboembolic Pulmonary Hypertension, CTEPH). Patients with CTEPH are diagnosed as inoperable. The investigators perform diagnostic tests on blood samples collected directly from the pulmonary artery during the right heart catheterization performed as part of the patients' routine medical care for the diagnosis of the disease or for follow-up 6 months after the initiation of PH-specific treatment. All blood samples are processed by platelet function analyzer-100 (PFA-100), light transmission aggregometry (LTA), rotational thromboelastometry (ROTEM) and endogenous thrombin potential (ETP).The primary objective of the study is to assess platelet function, coagulation and anti-coagulation pathways and fibrinolysis in PAH and inoperable CTEPH patients and to investigate the possible effects of PH- specific therapy on hemostasis.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary Arterial Hypertension,
* Chronic Thromboembolic Pulmonary Hypertension.

Exclusion Criteria:

* renal insufficiency,
* hepatic insufficiency,
* thyroid dysfunction,
* malignancy,
* active infections,
* receiving anticoagulant or antiplatelet therapy,
* history of hemostatic disorders irrelevant to their primary disease,
* abnormal red blood counts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study participants are recruited among the pulmonary hypertension patients of the Pulmonary Hypertension Unit, In the Second Department of Critical Care Medicine, Attiko University Hospital, Athens, Greece
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-03-12 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
PFA-100 in detection of platelet abnormalities in PAH and CTEPH patients. | 6 months
  Change in the percentage of PAH and CTEPH patients who are detected with platelet abnormalities in PFA-100 testing from the date of the first right heart catheterization performed for the diagnosis of their disease (before treatment implementation) to the date of the second right heart catheterization performed for follow-up (after treatment implementation) at 6 months.
Light transmission aggreggometry in detection of platelet abnormalities in PAH and CTEPH patients. | 6 months
  Change in the percentage of PAH and CTEPH patients who are detected with platelet abnormalities in LTA testing from the date of the first right heart catheterization performed for the diagnosis of their disease (before treatment implementation) to the date of the second right heart catheterization performed for follow-up (after treatment implementation) at 6 months.
ROTEM in detection of coagulation abnormalities in PAH and CTEPH patients. | 6 months
  Change in the percentage of PAH and CTEPH patients who are detected with coagulation abnormalities in ROTEM testing from the date of the first right heart catheterization performed for the diagnosis of their disease (before treatment implementation) to the date of the second right heart catheterization performed for follow-up (after treatment implementation) at 6 months.
Endogenous thrombin potential in detection of thrombin abnormalities in PAH and CTEPH patients. | 6 months
  Change in the percentage of PAH and CTEPH patients who are detected with thrombin deficits in endogenous thrombin potential testing from the date of the first right heart catheterization performed for the diagnosis of their disease (before treatment implementation) to the date of the second right heart catheterization performed for follow-up (after treatment implementation) at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Vrigkou, MD, MSc, Principal Investigator — National and Kapodistrian University of Athens; Argyrios Tsantes, MD, PhD, Study Director — National and Kapodistrian University of Athens; Iraklis Tsagkaris, MD, PhD, Study Chair — National and Kapodistrian University of Athens; Apostolos Armaganidis, MD, PhD, Study Chair — National and Kapodistrian University of Athens
Locations (1):
- Attikon University Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berger G, Azzam ZS, Hoffman R, Yigla M. Coagulation and anticoagulation in pulmonary arterial hypertension. Isr Med Assoc J. 2009 Jun;11(6):376-9. PMID 19697592
- [Background] Herve P, Humbert M, Sitbon O, Parent F, Nunes H, Legal C, Garcia G, Simonneau G. Pathobiology of pulmonary hypertension. The role of platelets and thrombosis. Clin Chest Med. 2001 Sep;22(3):451-8. doi: 10.1016/s0272-5231(05)70283-5. PMID 11590840
- [Background] Lopes AA, Caramuru LH, Maeda NY. Endothelial dysfunction associated with chronic intravascular coagulation in secondary pulmonary hypertension. Clin Appl Thromb Hemost. 2002 Oct;8(4):353-8. doi: 10.1177/107602960200800407. PMID 12516685
- [Background] Preston IR, Farber HW. Anti-coagulation in pulmonary arterial hypertension: the real blood and guts. J Thorac Dis. 2016 Sep;8(9):E1106-E1107. doi: 10.21037/jtd.2016.08.48. No abstract available. PMID 27747077
- [Background] Remkova A, Simkova I, Valkovicova T. Platelet abnormalities in chronic thromboembolic pulmonary hypertension. Int J Clin Exp Med. 2015 Jun 15;8(6):9700-7. eCollection 2015. PMID 26309645
- [Background] Lang IM, Dorfmuller P, Vonk Noordegraaf A. The Pathobiology of Chronic Thromboembolic Pulmonary Hypertension. Ann Am Thorac Soc. 2016 Jul;13 Suppl 3:S215-21. doi: 10.1513/AnnalsATS.201509-620AS. PMID 27571003